CLINICAL TRIAL: NCT06101394
Title: Study Protocol for Near-infrared Molecular Imaging for Lung Cancer Detection and Treatment During Mini-invasive Surgery (Phase II Trial) - (the RECOGNISE Study)
Brief Title: Development of a Fluorescent Visualization System for Non-visible Lung Cancer Nodules
Acronym: RECOGNISE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Turin, Italy (Other)
Collaborators: A.O.U. Città della Salute e della Scienza (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23537
Record Dates: First submitted 2023-03-27; First posted 2023-10-26 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Lung Cancer; Video-assisted Thoracic Surgery; EGFR; Cetuximab
MeSH Terms: conditions — Lung Neoplasms | interventions — Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- cetuximab-IRDye800 (Experimental): Infusion of the study drug will be performed 2-5 days before the surgery: the patients will receive 100 mg of cetuximab intravenously over 30 minutes and a dose 50 mg of cetuximab IRDye800 over 30 minutes to 1 hour.
  Interventions: Drug: Cetuximab-IRDye800

INTERVENTIONS:
Drug: Cetuximab-IRDye800 — Infusion of the study drug will be performed 2-5 days before the surgery: the patients will receive 100 mg of cetuximab intravenously over 30 minutes and a dose 50 mg of cetuximab-IRDye800 over 30 minutes to 1 hour.
  Other Names: Cetuximab

SUMMARY:
To date, lung resection and lymphadenectomy remain the best curative option in patients with early-stage non-small cell lung cancer. Moreover, cancer screening programs have led to a frequent diagnoses of indeterminate lung lesions, many of which require surgical biopsy for diagnosis and intervention. Additionally, pre-operative imaging assessment frequently underestimates lymph-node involvement. Finally, the increase in the utilization of minimally invasive procedures remains mandatory.

The aim of our project is to verify if Cetuximab-IRDye800 could detect cancer nodules and lymph node metastases during minimally invasive thoracic surgery. A result favoring the use of Cetuximab-IRDye800 would permit the use of a minimally invasive approach to a more significant number of patients, which are presently operable only by a traditional "open" approach. Consequentially, it would lead to an improvement in surgical outcomes, a reduction of costs, and an enhanced patient quality of life.

In addition, a result favoring Cetuximab-IRDye800 could consent to correctly remove mislead metastatic lymph nodes (i.e., unexpected lymph-nodes metastasis) and neoplastic localization unidentified at pre-operative diagnostic assessments. It would lead to more accurate cancer staging, and a tailored post-operative treatment. Finally, the investigators expect to validate using Cetuximab-IRDye800 as an optimal tracker that can be easily applied intraoperatively during minimally invasive surgical procedures.

DETAILED DESCRIPTION:
Lung cancer is the leading cause of cancer deaths in the European Union (EU) (267,000 deaths/year) and the fourth most common cancer (321,000 new cases/year). To date, radical surgery remains the best curative option in patients with early-stage lung cancer. Moreover, cancer screening programs have led to frequent diagnoses of indeterminate lung lesions, many requiring surgical biopsy for diagnosis and intervention.

For example, available data showed that 5.9 % of the European population over 15 years of age consumed at least 20 cigarettes per day (8.4 % in the male population), and around 12.6 % consumed less than 20. The recent lung cancer screening studies documented a prevalence of indeterminate pulmonary nodules as high as 50% in high-risk smokers, with a cancer detection rate in the overall screened population of 1%. Fascinatingly, 69% of screen-detected lung cancers were detected at early stage IA or IB.

Finally, studies on lung cancer screening, like the NELSON trial, showed a 26% reduction in lung cancer deaths at 10 years. The potential social impact of the present project is linked to establishing this screening program in Europe. One could estimate that if applied in the high-risk European population (i.e., high smokers), the screening could identify 3.5 million indeterminate pulmonary nodules, of which 250,000 are early-stage lung cancer. [2] Therefore, using the NIR-tracker the investigators propose could consent to a minimally invasive surgery in this scenario as a diagnostic and therapeutic procedure. Consequently, it could determine the reduction of time to diagnosis, morbidity, mortality, and costs of postoperative care associated with more invasive surgical procedures.

To date, lung anatomical resection with lymphadenectomy remains the best curative option in patients with early-stage non-small cell lung cancer. Moreover, cancer screening programs have led to frequent diagnoses of indeterminate lungs, many requiring surgical biopsy for diagnosis and intervention.

Nevertheless, the increase in the utilization of minimally invasive procedures (e.g., video-assisted thoracic surgery -VATS- and robotic-assisted thoracic surgery -RATS- ) remains mandatory in order to reduce the significant morbidity of classic surgery, the surgical trauma, to preserve organs function and to improve patient's quality of life. Nevertheless, minimally invasive surgery represents the surgical approach of choice in less than 40% of lung anatomical resections conducted in Europe. One of the significant issues that hinder the application of VATS and RATS to most early-stage NSCLC patients is the difficulty of recognizing lung nodules located deep in the lung parenchyma and, consequently, not visible with the traditional camera system. Indeed, VATS and RATS do not consent to manual lung palpation, making localizing the not superficial lung nodule problematic.

Several approaches have been developed to enhance the localization of indeterminate lung nodules and decrease the time to diagnosis and rate of conversion to open surgery. Nevertheless, none of these is 100% sensitive or without complications, also of severe grade.

Numerous pre-operative methods are being employed, including percutaneous CT-guided placement techniques, encompassing the use of microcoils, hook-wires, and spiral-wires. These devices can support nodule localization during minimally invasive lung procedures; nevertheless, they could be easily displaced during patient transport and positioning, intraoperative atelectasis, single lung ventilation, and surgeon manipulation. Moreover, some locations of the lung as the apex, near the diaphragm, and the proximity of mediastinum and great vessels. Furthermore, all these pre-operative localization techniques require two different procedures, one for the CT-guided referral placement and one for surgical treatment. Finally, the rate of pneumothorax, hemorrhage, and subcutaneous emphysema are not insignificant, and these complications are mandatory to avoid in several sub-groups of patients. Other pre-operative methods encompass the use of dye marking by methylene blue or fluorescent. [8] Nevertheless, the accuracy of the staining of the targeted area is greatly affected by the time between tumor marking and thoracoscopy. In particular, the significant impact is on the difficulty in dye visualization during operation, limited information on lesion depth, and rapid diffusion of dye into surrounding lung parenchyma between the time of injection and surgery. Of note, methylene blue has limited application in patients with anthracotic pigmentation. Moreover, also these techniques require two procedures for diagnosis and treatment. Lastly, these procedures remain complicated by the risk of pneumothorax, hemorrhage, dye air embolism, and cerebrovascular accident, and cases of lethal anaphylaxis to the dye of choice.

On the other hand, clinical pre-operative staging and surgical planning are based on pre-operative images taken before surgery, either by computed tomography (CT), positron emission tomography (PET), or magnetic resonance imaging (MRI). These pre-operative imaging assessments frequently underestimate lymph node involvement and secondary localizations. This results in an upstaging after surgical resection ranging from 9 to 24 % in clinical Stage I lung cancer. [10, 11] Nevertheless, the current system of intraoperative imaging, based on direct injection of a tracker in the principal tumoral mass, demonstrated a substantial limitation in lung cancer. This is principally due to the deeper location of the lymph node, usually profoundly engaged in normal fat tissue, and to the irregular lymph node drain system in the respiratory region.

In this context, intraoperative fluorescence imaging can enhance the real-time identification of cancer cells during minimally invasive surgical procedures. This could overcome the difficulty of finding cancer nodules located deep in the lung parenchyma, not visible on the surface of normal, uninvolved tissue. The Near-infrared (NIR) fluorescence (700-1,000 nm) detection avoids the natural background fluorescence interference of biomolecules, which provides high contrast between the target and background tissues in small animals. NIR fluorophores have a more comprehensive dynamic range and minimal background fluorescence because of reduced scattering compared with visible fluorescence detection. However, the conventional near-infrared (NIR) indocyanine green (ICG) method demonstrated a significant limitation in deep cancer recognition, principally due to its intrinsic low-depth tissue penetration. Similarly, the lymph-node sentinel approach conducted by the ICG method proved to be inefficient, mainly due to the non-specificity of the tracker and the irregular pathway of pulmonary lymph node drainage.

The IRDye® 800CW is an indocyanine-type NIR fluorophore with peak absorption at 775 nm and peak excitation emission at 796 nm. It provides a quantum yield of 9% with an extinction coefficient of 242,000 M-1cm-1. It has a molecular weight of 962 Da. The IRDye® 800CW demonstrated enhanced tissue penetration compared to other NIR dyes.

Epidermal growth factor (EGF) is a 53-amino acid cytokine (6.2 kDa) that is secreted by ectodermic cells, monocytes, kidneys, and duodenal glands. EGF stimulates the growth of epidermal and epithelial cells. EGF and at least seven other growth factors and their transmembrane receptor kinases play essential roles in cell proliferation, invasion, metastasis, neovascularization, adhesion, migration, differentiation, and inhibition of apoptosis. The EGF receptor (EGFR) family consists of four transmembrane receptors, which include EGFR (HER1/erbB-1), HER2 (erbB-2/neu), HER3 (erbB-3), and HER4 (erbB-4); and is commonly overexpressed in lung cancer. Cetuximab is a monoclonal antibody able to inhibit and degrade the EGFR. Given by intravenous infusion (IV), Cetuximab binds to the EGFR and stops the binding and activation of the downstream signaling pathways. Moreover, as the investigators previously published, EGFR mutation is linked with skip-metastasis phenomena (i.e., pathologically proved mediastinal lymph node involvement in the absence of intrapulmonary or hilar lymph node disease).

The combination with the clinical approved monoclonal antibody anti-epidermal growth factor EGFR Cetuximab (Cetuximab-IRDye800) has shown promising results as a specific tracker in other cancer types (i.e., brain, pancreas, head, and neck). The investigators hypothesize that using Cetuximab-IRDye800 during minimally invasive surgical procedures for lung cancer could overcome the limitation demonstrated by ICG and the traditional localization strategies (e.g., coil, hook, dye intra-tumoral injection). The investigators expect to validate using an optimal tracker that can be easily applied intraoperatively during minimally invasive lung surgical procedures. The investigators expect to define the optimal time window and the optimal dose of administration of the tracker. The investigators expect to discover neoplastic localization in lymph nodes and lung parenchyma not predictable pre-operatively.

ELIGIBILITY:
Inclusion criteria:

1. Clinical Stage I non-small cell lung cancer
2. - Considered candidate to minimally invasive surgical resection after pre-operative assessment
3. Adequate organ function
4. Performance status (ECOG) ≤2
5. Potentially fertile female subjects must agree to use highly effective contraception throughout the - study and for three months after the last dose of the study medication
6. Written informed consent

Exclusion criteria:

1. Previous systemic treatments for lung cancer
2. Previous radiotherapy on lung or mediastinum
3. - Concomitant disorders that compromise the ability to adhere to the procedures of the Protocol
4. Hemoglobin < 9 gm/dL
5. Platelet count < 100,000/mm³
6. Leukocyte count < 3000/mm³
7. Absolute neutrophil count < 1500/mm³
8. Magnesium, potassium, and calcium < the lower limit of normal per institution normal lab values
9. Thyroid-stimulating hormone (TSH) > 13 micro international units/mL
10. Received an investigational drug within 30 days or 5 half-life prior to the first dose of cetuximab IRDye800
11. Within 6 months prior to enrollment, myocardial infarction; cerebrovascular accident; uncontrolled congestive heart failure; significant liver disease; or unstable angina
12. History of infusion reactions to cetuximab or other monoclonal antibody therapies
13. Evidence of QT prolongation on pretreatment electrocardiogram (ECG) (greater than 440 ms in males or greater than 450 ms in females)
14. Hypersensitivity to Cetuximab-IRDye800, Cetuximab, or any of the excipients.
15. Receiving class IA (quinidine, procainamide) or class III (dofetilide, amiodarone, sotalol) antiarrhythmic agents
16. Pregnancy, assessed by a pregnancy serum test (βhCG), or breastfeeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Nodule Detection | The detection of lung nodules' NIR emission was registered in the first 5 minutes of the NIR camera activation during surgery.
  The proportion of patients with detection of lung nodules during surgery by NIR camera, with respect to the pathology report.

SECONDARY OUTCOMES:
Lymph node detection | The lymph-nodal NIR emission was revealed and registered during surgery at the same time as the lymph-nodal dissection was performed.
  The proportion of patients with detection of lymph nodal metastatic disease during surgery by NIR camera, with respect to the pathology report.
Unexpected cancer localization detection | Unexpected localization of NIR emission was researched and registered at the end of standard surgical procedure with systematic research of 10 minutes.
  The proportion of patients with detection of unexpected cancer localization during surgery by NIR camera, with respect to the pathology report.
Negative surgical margins, with respect to the pathology report. | The nature of the surgical margin (e.g., if neoplastic or not) will be registered during pathological examination of the specimen, up to 15 days after surgical procedure
  The proportion of patients with negative surgical margins, with respect to the pathology report.
Detection speed | The detection time of NIR emission was registered in the first 5 minutes of activation of the NIR camera, at the beginning of surgical procedure, after all the pleurotomy have been performed.
  Time spawns between the insertion of the NIR camera and the visualization of the nodule. Localization of the fluorescent compound in the known nodule will be annotated.
Toxicity Incidence | The morbidity or toxicity will be assessed during and after drug infusion (Day0), during and after a hospital stay (Day1 to Day13), and during the control visits (in averange until the first year after drug infusion).
  Toxicity will be recorded and classified according to the definitions of the NCI criteria "Common Terminology Criteria for Adverse Events (CTCAE)", version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Enrico Ruffini, M.D., Study Director — Department of Surgical Science, University of Torino, Torino, Italy; Francesco Guerrera, M.D., Ph.D., Principal Investigator — Department of Surgical Science, University of Torino, Torino, Italy
Locations (2):
- Italy (2):
  - Azienda Ospedaliera Universitaria Città della Salute e della Scienza di Torino, Torino, TO
  - S.C. Chirurgia Toracica U, Città della Salute e della Scienza di Torino, Torino

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Beffa ED, Lyberis P, Rosboch GL, Arezzo A, Lococo F, Carena L, Sciorsci E, Monica V, Lausi PO, Dusi V, Busardo FP, Buffa E, Stefania R, Ciccone G, Monagheddu C, Capello BM, Vancheri R, Garrone P, Gabbarini F, Cattel F, Ruffini E, Guerrera F. Study protocol for Near-infrared molecular imaging for lung cancer detection and treatment during mini-invasive surgery (phase II Trial) - (the RECOGNISE study). BMC Cancer. 2024 Sep 2;24(1):1078. doi: 10.1186/s12885-024-12859-6. PMID 39218855